CLINICAL TRIAL: NCT01754155
Title: A Prospective Radiostereometric Analysis and Clinical Evaluation of the Zimmer® Continuum® Acetabular Cup With Vitamin E Stabilized Polyethylene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central DuPage Hospital (Other)
Collaborators: Zimmer Biomet (Industry); Halifax Biomedical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CW55584
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Radiostereometric Analysis; Vitamin E Liner; Zimmer® Continuum® Acetabular Cup
Keywords: Vitamin E; Zimmer; RSA; Radiostereometric Analysis

ARMS (1):
- Vitamin E Polyethylene and RSA (Other): All subjects will have the Vitamin E polyethylene and RSA beads placed during surgery. Subjects will then have standard x-ray images and RSA images taken at specific time points up until 2 years post-operatively.
  Interventions: Radiation: RSA images

INTERVENTIONS:
Radiation: RSA images — All subjects will have the Vitamin E polyethylene and RSA beads placed during surgery. Subjects will then have standard x-ray images and RSA images taken at specific time points up until 2 years post-operatively.

SUMMARY:
The purpose of this study is to use Radiostereometric Analysis (RSA) and clinical outcome measures to evaluate early, post-operative implant stability, post-operative implant fixation, clinical performance, and in-vivo wear of the Zimmer® Continuum® Cup with vitamin E stabilized polyethylene.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the hip indicating surgical intervention
* Scheduled to undergo an uncemented total hip arthroplasty (THA)
* Patients between the ages of 18 and 65, inclusive
* Ability to give informed consent
* Patients will be available for follow-up for a minimum of 2 years after surgery

Exclusion Criteria:

* Patients less than 18 years of age, or older than 65 years of age.
* Post-traumatic arthritis in the affected hip
* Rheumatoid arthritis in the affected hip
* Hip dysplasia in the affected hip
* Prior arthroplasty of the affected hip
* Active or prior infection of the affected hip
* Morbid obesity (BMI > 35)
* Medical condition precluding major surgery
* Severe osteoporosis or osteopenia
* Neuromuscular impairment
* Patients with known allergy to metals
* Pregnancy
* Patients with compromised kidney function
* Patient is immuno-suppressed
* Patients that require a femoral head less than 32 mm or greater than 40mm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Assessing the Continuum® Cup for adequate fixation to the underlying bone as measured by migration and tilt | 2 years
Assessing the migration pattern of the Continuum® Cup | 2 years
Determining a correlation between radiolucent lines (RLLs) measured by Charnley-DeLee Zone Analyses and migration characteristics using RSA | 2 years
Determine if inducible displacement is indicative of adequate fixation | 2 years
Assess the health status and functional outcome of patients with the Continuum® Cup | 2 years
Assess the wear rate of the Vitamin E polyethylene with a ceramic femoral head | 2 years
Determine if the wear rate of the Vitamin E liner is the same in-vivo as it is in simulation testing | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott Sporer, MD, Principal Investigator — Central DuPage Hospital
Locations (1):
- Central DuPage Hospital, Winfield, Illinois, United States